CLINICAL TRIAL: NCT00005442
Title: Re-evaluating Triglycerides in Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4371; R29HL051024 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertriglyceridemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertriglyceridemia

SUMMARY:
To conduct a comprehensive epidemiologic investigation into the relationship between serum triglyceride (TG) levels and coronary heart disease (CHD).

DETAILED DESCRIPTION:
BACKGROUND:

The results of this investigation helped to shed substantial light on the controversial relationship between triglycerides and coronary heart disease, a topic of great importance to preventive cardiology. Additionally, important methodological information was obtained in the study of interactions and precision of variables in epidemiologic analysis.

DESIGN NARRATIVE:

There were three components to the study: 1) an analysis of several existing cardiovascular databases for evidence of a significant association between coronary heart disease and specific lipid interactions involving triglycerides; 2) an analysis of these databases to investigate the role of measurement precision on the association between elevated triglyceride levels and coronary heart disease; and 3) a survey of both expert lipidologists and community clinicians to examine current practices related to screening for and treatment of elevated triglyceride levels for the purpose of reducing coronary heart disease risk. Five databases were used in the first two components of this study. These data sets included those of the Lipid Research Clinics Prevalence and Mortality Follow-up Studies; the Lipid Research Clinics Coronary Primary Prevention Trial; the Multiple Risk Factor Intervention Trial; the National Heart, Lung, and Blood Type II Coronary Intervention Study; and the Coronary Drug Project. For the first component, detailed statistical analyses of all databases were performed, specifically examining the role of lipid interactions involving triglycerides and their association with coronary heart disease. For the second component, more precise estimates of each subject's lipid levels were recalculated using the multiple lipid measurements already available in each database. Each dataset was then analyzed for evidence of an independent relationship between triglycerides and coronary heart disease and to validate the theoretical findings suggesting that measurement imprecision may explain the difficulty of detecting an independent triglyceride-coronary heart disease association. The public health implications of the current state of knowledge surrounding triglycerides were assessed with survey research techniques in the third component.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1994-06; Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Avins — University of California at San Francisco

REFERENCES:
- [Background] Avins AL, Browner WS. Lowering risk without lowering cholesterol: implications for national cholesterol policy. Ann Intern Med. 1996 Sep 15;125(6):502-6. doi: 10.7326/0003-4819-125-6-199609150-00012. PMID 8779464
- [Background] Avins AL, Browner WS. Improving the prediction of coronary heart disease to aid in the management of high cholesterol levels: what a difference a decade makes. JAMA. 1998 Feb 11;279(6):445-9. doi: 10.1001/jama.279.6.445. PMID 9466637
- [Background] Avins AL, Neuhaus JM. Do triglycerides provide meaningful information about heart disease risk? Arch Intern Med. 2000 Jul 10;160(13):1937-44. doi: 10.1001/archinte.160.13.1937. PMID 10888968